CLINICAL TRIAL: NCT01134263
Title: Lot-to-Lot Consistency and Bridging Study of a Tetravalent Dengue Vaccine in Healthy Adults in Australia
Brief Title: Study of a Tetravalent Dengue Vaccine in Healthy Adults in Australia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CYD17; U1111-1114-7646 (Other: WHO)
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-05

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue Fever; Dengue Hemorrhagic Fever; CYD Dengue Vaccine; Lot Consistency
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: An observer-blind procedure was followed for the three injections with CYD dengue vaccine or placebo. Neither the observer, Investigator, Sponsor, nor the participant knew which product was administered.
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- CYD Dengue Vaccine Phase III Lot 1 (Experimental): Participants received 3 doses of CYD dengue vaccine (Phase III Lot 1), one each at Day 0 (vaccination 1),Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
  Interventions: Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, & 4 virus
- CYD Dengue vaccine - Phase III Lot 2 (Experimental): Participants received 3 doses of CYD dengue vaccine (Phase III Lot 2) one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
  Interventions: Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, & 4 virus
- CYD Dengue vaccine - Phase III Lot 3 (Experimental): Participants received 3 doses of CYD dengue vaccine (Phase III Lot 3) one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
  Interventions: Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, & 4 virus
- CYD Dengue vaccine - Phase II Lot (Experimental): Participants received 3 doses of CYD dengue vaccine (Phase II Lot) one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
  Interventions: Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, & 4 virus
- Placebo (Placebo Comparator): Participants received placebo matched to CYD dengue vaccine, one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
  Interventions: Biological: Placebo: NaCl 0.9%

INTERVENTIONS:
Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, & 4 virus — 0.5 ml, Subcutaneous (SC)
  Other Names: CYD Dengue vaccine
  Arms: CYD Dengue Vaccine Phase III Lot 1
Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, & 4 virus — 0.5 ml, SC
  Other Names: CYD Dengue vaccine
  Arms: CYD Dengue vaccine - Phase III Lot 2
Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, & 4 virus — 0.5 ml, SC
  Other Names: CYD Dengue vaccine
  Arms: CYD Dengue vaccine - Phase III Lot 3
Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, & 4 virus — 0.5 ml, Subcutaneous (SC)
  Other Names: CYD Dengue vaccine
  Arms: CYD Dengue vaccine - Phase II Lot
Biological: Placebo: NaCl 0.9% — 0.5 ml, SC
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
The purpose of this study was to demonstrate that different CYD dengue vaccine lots manufactured using the same method and in the same location but at different times produce an equivalent immunological response after 3 doses.

Primary Objective

* To demonstrate that three different Phase III lots of CYD dengue vaccine induce an equivalent immune response in terms of post-Dose 3 geometric mean titers (GMTs) against the four parental serotypes.

Secondary Objectives:

* To demonstrate that data from one Phase II lot and pooled data from Phase III lots of CYD dengue vaccine show an equivalent immune response in terms of post-Dose 3 GMTs against the four parental serotypes.
* To describe the safety of the CYD dengue vaccine in all participants after each dose.

DETAILED DESCRIPTION:
All participants received 3 doses of their assigned vaccine or placebo and provided blood samples at defined timepoints for flavivirus status and immunogenicity assessment. Safety data were collected in all participants after each dose and throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years on the day of inclusion.
* Informed consent form was signed and dated.
* Able to attend all scheduled visits and to comply with all trial procedures.
* For a woman of childbearing potential, use of an effective method of contraception, or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination (i.e., for 14 months).

Exclusion Criteria:

* Known pregnancy, or a positive urine pregnancy test.
* History of flavivirus infection or vaccination or prolonged habitation in a dengue endemic area.
* Currently breastfeeding a child.
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination, except for pandemic influenza vaccination.
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Self-reported seropositivity for human immunodeficiency virus (HIV).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Identified as a site employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the site employees or the Investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 715 (Actual)
Dates: Start 2010-10-05 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (7):
- Australia (7):
  - Adelaide
  - Carina Heights
  - Enoggera
  - Heidelberg
  - Herston
  - Subiaco
  - Westmead

REFERENCES:
- [Result] Torresi J, Heron LG, Qiao M, Marjason J, Chambonneau L, Bouckenooghe A, Boaz M, van der Vliet D, Wallace D, Hutagalung Y, Nissen MD, Richmond PC. Lot-to-lot consistency of a tetravalent dengue vaccine in healthy adults in Australia: a randomised study. Vaccine. 2015 Sep 22;33(39):5127-34. doi: 10.1016/j.vaccine.2015.08.008. Epub 2015 Aug 13. PMID 26279339
- [Derived] Torresi J, Richmond PC, Heron LG, Qiao M, Marjason J, Starr-Spires L, van der Vliet D, Jin J, Wartel TA, Bouckenooghe A. Replication and Excretion of the Live Attenuated Tetravalent Dengue Vaccine CYD-TDV in a Flavivirus-Naive Adult Population: Assessment of Vaccine Viremia and Virus Shedding. J Infect Dis. 2017 Oct 17;216(7):834-841. doi: 10.1093/infdis/jix314. PMID 28968794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 05 October 2010 to 26 November 2010 at 8 study sites in Australia.
Pre-assignment Details: A total of 715 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled in the study.
Groups:
- CYD Dengue Vaccine Phase III Lot 1: Participants received 3 doses of CYD dengue vaccine (Phase III Lot 1), one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
- CYD Dengue Vaccine Phase III Lot 2: Participants received 3 doses of CYD dengue vaccine (Phase III Lot 2) one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
- CYD Dengue Vaccine Phase III Lot 3: Participants received 3 doses of CYD dengue vaccine (Phase III Lot 3) one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
- CYD Dengue Vaccine Phase II Lot: Participants received 3 doses of CYD dengue vaccine (Phase II Lot) one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Phase III Lot 1 | CYD Dengue Vaccine Phase III Lot 2 | CYD Dengue Vaccine Phase III Lot 3 | CYD Dengue Vaccine Phase II Lot | Placebo
Started | 164 | 163 | 163 | 168 | 57
Received Vaccination 1 | 163 | 162 | 163 | 167 | 57
Received Vaccination 2 | 151 | 152 | 139 | 154 | 53
Received Vaccination 3 | 140 | 145 | 134 | 151 | 49
Safety Population (Safety Population:All participants who received study drug, analyzed according to treatment received) | 163 | 161 | 164 (1 participant randomized to the Phase III Lot 2 group, received Phase III Lot 3 vaccination.) | 167 | 57
Completed | 140 | 143 | 134 | 149 | 48
Not Completed | 24 | 20 | 29 | 19 | 9
Not completed — Serious adverse event | 2 | 1 | 1 | 1 | 1
Not completed — Other adverse event | 1 | 2 | 5 | 3 | 0
Not completed — Protocol Violation | 8 | 7 | 2 | 4 | 2
Not completed — Lost to Follow-up | 4 | 3 | 5 | 3 | 1
Not completed — Withdrawal by Subject | 8 | 6 | 16 | 7 | 5
Not completed — Enrolled, but not treated | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Full Analysis Set included all participants who received at least 1 injection of CYD Dengue Vaccine or placebo.
Groups:
- CYD Dengue Vaccine Phase III Lot 3: Participants received 3 doses of 0.5 ml CYD dengue vaccine (Phase III Lot 3) one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
- CYD Dengue Vaccine Phase II Lot: Participants received 3 doses of 0.5 ml CYD dengue vaccine (Phase II Lot) one each at Day 0 (vaccination 1), 6 (vaccination 2), and 12 (vaccination 3) months, subcutaneously.
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Phase III Lot 1 | CYD Dengue Vaccine Phase III Lot 2 | CYD Dengue Vaccine Phase III Lot 3 | CYD Dengue Vaccine Phase II Lot | Placebo | Total
Number analyzed (Participants) | 163 | 162 | 163 | 167 | 57 | 712
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.4 (13.3) | 39.4 (12.9) | 38.7 (14.1) | 38.4 (13.2) | 39.7 (13.5) | 39.0 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 87 | 84 | 84 | 33 | 391
  Male | 60 | 75 | 79 | 83 | 24 | 321

OUTCOME MEASURES:

1. Primary Outcome: Post-Dose 3 Geometric Mean Titers (GMTs) of Antibodies Against Each of the Four Dengue Virus Serotypes Following Vaccination With Phase III Lots of CYD Dengue Vaccine
Description: GMTs against each of the 4 serotypes (serotype 1, serotype 2, serotype 3 and serotype 4) of dengue virus strains were assessed using the plaque reduction neutralization test (PRNT) assay. The lot-to-lot consistency between 3 Phase III lots was based on the use of the two-sided 95% confidence interval (CI) of the differences of the means of the log10 transformed post-vaccination titers between pairs of lots.
Time Frame: 28 days post-injection 3
Population: Analysis was performed on Per-protocol analysis set which included participants who received at least 1 dose of the study vaccine or placebo and had no protocol deviations. Data for this outcome measure was not planned to be collected and analyzed for Phase II Lot and placebo.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Groups:
- CYD Dengue Vaccine Phase III Lot 2: Participants received 3 doses of CYD dengue vaccine (Phase III Lot 2) one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month12 (vaccination 3), subcutaneously.
- CYD Dengue Vaccine Phase III Lot 3: Participants received 3 doses of CYD dengue vaccine (Phase III Lot 3) one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month12 (vaccination 3) , subcutaneously.
Arm/Group | CYD Dengue Vaccine Phase III Lot 1 | CYD Dengue Vaccine Phase III Lot 2 | CYD Dengue Vaccine Phase III Lot 3
Number analyzed (Participants) | 129 | 123 | 124
Titer (1/dilution)
  Dengue Virus Serotype 1 | 20.6 [16.9 to 25.1] | 18.1 [14.8 to 22.2] | 17.1 [13.9 to 21.2]
  Dengue Virus Serotype 2 | 65.9 [50.6 to 85.7] | 44.1 [33.3 to 58.3] | 58.1 [43.2 to 78.2]
  Dengue Virus Serotype 3 | 74.2 [60.1 to 91.7] | 65 [53.2 to 79.3] | 71.6 [58.2 to 88.2]
  Dengue Virus Serotype 4 | 131.8 [101.4 to 171.3] | 94.6 [75.3 to 118.7] | 108.5 [84.2 to 139.7]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Phase III Lot 1 vs CYD Dengue Vaccine Phase III Lot 2; Dengue Virus Serotype 1: Phase III Lot 1 vs Lot 2; Test type: Equivalence — Lot consistency for each pair of lots was demonstrated if, for each pair of lots and each serotype the lower limit of the 95% CI was > -0.301 and the upper limit was < 0.301; Difference of Log10 GMT = 0.055, 95% CI 2-sided [-0.067 to 0.178]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Phase III Lot 2 vs CYD Dengue Vaccine Phase III Lot 3; Dengue Virus Serotype 1: Phase III Lot 2 vs Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Log10 GMT = 0.024, 95% CI 2-sided [-0.102 to 0.151]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine Phase III Lot 1 vs CYD Dengue Vaccine Phase III Lot 3; Dengue Virus Serotype 1: Phase III Lot 3 vs Lot 1; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Log10 GMT = -0.080, 95% CI 2-sided [-0.204 to 0.045]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine Phase III Lot 1 vs CYD Dengue Vaccine Phase III Lot 2; Dengue Virus Serotype 2: Phase III Lot 1 vs Lot 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Log10 GMT = 0.174, 95% CI 2-sided [0.009 to 0.340]
Statistical Analysis 5: Comparison: CYD Dengue Vaccine Phase III Lot 2 vs CYD Dengue Vaccine Phase III Lot 3; Dengue Virus Serotype 2: Phase III Lot 2 vs Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Log10 GMT = -0.120, 95% CI 2-sided [-0.297 to 0.056]
Statistical Analysis 6: Comparison: CYD Dengue Vaccine Phase III Lot 1 vs CYD Dengue Vaccine Phase III Lot 3; Dengue Virus Serotype 2: Phase III Lot 3 vs Lot 1; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Log10 GMT = -0.054, 95% CI 2-sided [-0.225 to 0.117]
Statistical Analysis 7: Comparison: CYD Dengue Vaccine Phase III Lot 1 vs CYD Dengue Vaccine Phase III Lot 2; Dengue Virus Serotype 3: Phase III Lot 1 vs Lot 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Log10 GMT = 0.058, 95% CI 2-sided [-0.068 to 0.184]
Statistical Analysis 8: Comparison: CYD Dengue Vaccine Phase III Lot 2 vs CYD Dengue Vaccine Phase III Lot 3; Dengue Virus Serotype 3: Phase III Lot 2 vs Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Log10 GMT = -0.042, 95% CI 2-sided [-0.167 to 0.082]
Statistical Analysis 9: Comparison: CYD Dengue Vaccine Phase III Lot 1 vs CYD Dengue Vaccine Phase III Lot 3; Dengue Virus Serotype 3: Phase III Lot 3 vs Lot 1; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Log10 GMT = -0.016, 95% CI 2-sided [-0.144 to 0.113]
Statistical Analysis 10: Comparison: CYD Dengue Vaccine Phase III Lot 1 vs CYD Dengue Vaccine Phase III Lot 2; Dengue Virus Serotype 4: Phase III Lot 1 vs Lot 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Log10 GMT = 0.144, 95% CI 2-sided [-0.006 to 0.295]
Statistical Analysis 11: Comparison: CYD Dengue Vaccine Phase III Lot 2 vs CYD Dengue Vaccine Phase III Lot 3; Dengue Virus Serotype 4: Phase III Lot 2 vs Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Log10 GMT = -0.060, 95% CI 2-sided [-0.207 to 0.088]
Statistical Analysis 12: Comparison: CYD Dengue Vaccine Phase III Lot 1 vs CYD Dengue Vaccine Phase III Lot 3; Dengue Virus Serotype 4: Phase III Lot 3 vs Lot 1; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Log10 GMT = -0.085, 95% CI 2-sided [-0.242 to 0.073]

2. Secondary Outcome: Geometric Mean Titers of Antibodies Against Each of the Four Dengue Virus Serotypes Following Vaccination With Pooled Phase III Lots (1, 2 or 3 )and Phase II Lot of CYD Dengue Vaccine
Description: GMTs against each of the 4 serotypes (serotype 1, serotype 2, serotype 3 and serotype 4) of dengue virus strains were assessed using PRNT assay. Equivalence of Phase III vaccine with Phase II vaccine was assessed by Bridging between Phase III and Phase II Lot of CYD Dengue Vaccine.
Time Frame: 28 days post-Injection 3
Population: Analysis was performed on Per Protocol Analysis Set. Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for placebo.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Groups:
- CYD Dengue Vaccine Pooled Phase III Lot: Participants received 3 doses of CYD dengue vaccine one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3) from any of the Phase III Lots 1, 2 or 3.
Arm/Group | CYD Dengue Vaccine Pooled Phase III Lot | CYD Dengue Vaccine Phase II Lot
Number analyzed (Participants) | 376 | 128
Titer (1/dilution)
  Dengue Virus Serotype 1 | 18.6 [16.5 to 20.9] | 15.1 [12.4 to 18.4]
  Dengue Virus Serotype 2 | 55.4 [47.2 to 65.1] | 25.7 [20.6 to 32]
  Dengue Virus Serotype 3 | 70.2 [62.4 to 79.1] | 83.6 [71.1 to 98.4]
  Dengue Virus Serotype 4: number analyzed (Participants) | 376 | 127
  Dengue Virus Serotype 4 | 110.9 [96.1 to 127.9] | 115.4 [92.8 to 143.5]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Pooled Phase III Lot vs CYD Dengue Vaccine Phase II Lot; Dengue Virus Serotype 1; Test type: Equivalence — Equivalence between the pooled Phase III and Phase II was demonstrated if, for each serotype the lower limit of the 95%CI was > -0.301 and the upper limit was < 0.301; Difference of Log10 GMT = 0.091, 95% CI 2-sided [-0.009 to 0.192]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Pooled Phase III Lot vs CYD Dengue Vaccine Phase II Lot; Dengue Virus Serotype 2; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Difference of Log10 GMT = 0.334, 95% CI 2-sided [0.202 to 0.466]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine Pooled Phase III Lot vs CYD Dengue Vaccine Phase II Lot; Dengue Virus Serotype 3; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Difference of Log10 GMT = -0.076, 95% CI 2-sided [-0.173 to 0.021]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine Pooled Phase III Lot vs CYD Dengue Vaccine Phase II Lot; Dengue Virus Serotype 4; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Difference of Log10 GMT = -0.017, 95% CI 2-sided [-0.137 to 0.103]

3. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions After Any Vaccination
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Pain: Grade 3: Significant; prevents daily activity. Erythema and Swelling: Grade 3: > 10 cm. Participants with Injection Site Reactions of any Grade (1, 2 or 3) and grade 3 were reported.
Time Frame: 7 days post any vaccination
Population: Analysis was performed on Safety Analysis Set which included all participants who received the study dose, and participants were analyzed according to the treatment received. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Groups:
- CYD Dengue Vaccine Phase III Lot 1: Participants received 3 doses of 0.5 ml CYD dengue vaccine (Phase III Lot 1), one each at Day 0 (vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
Arm/Group | CYD Dengue Vaccine Phase III Lot 1 | CYD Dengue Vaccine Phase III Lot 2 | CYD Dengue Vaccine Phase III Lot 3 | CYD Dengue Vaccine Phase II Lot | Placebo
Number analyzed (Participants) | 163 | 161 | 164 | 167 | 57
Participants
  Pain: Any: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Pain: Any | 73 | 74 | 73 | 78 | 11
  Pain: Grade 3: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Pain: Grade 3 | 1 | 1 | 1 | 0 | 0
  Erythema: Any: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Erythema: Any | 22 | 15 | 25 | 24 | 0
  Erythema: Grade 3: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Erythema: Grade 3 | 0 | 0 | 0 | 0 | 0
  Swelling: Any: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Swelling: Any | 8 | 4 | 2 | 5 | 1
  Swelling: Grade 3: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Swelling: Grade 3 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Solicited Systemic Reactions After Any Vaccination
Description: Solicited systemic reactions: Asthenia, Fever, Headache, Malaise and Myalgia. Fever: Grade 3: >=39.0°C (>=102.1°F). Headache, malaise, myalgia and asthenia: Grade 3: significant; prevents daily activity. Participants with systemic reactions of any Grade (1, 2 or 3) and grade 3 were reported.
Time Frame: 14 days post any vaccination
Population: Analysis was performed on Safety Analysis Set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Groups:
- CYD Dengue Vaccine Phase II Lot: Participants received 3 doses of CYD dengue vaccine (Phase II Lot) one each at Day 0(vaccination 1), Month 6 (vaccination 2), and Month 12 (vaccination 3), subcutaneously.
Arm/Group | CYD Dengue Vaccine Phase III Lot 1 | CYD Dengue Vaccine Phase III Lot 2 | CYD Dengue Vaccine Phase III Lot 3 | CYD Dengue Vaccine Phase II Lot | Placebo
Number analyzed (Participants) | 163 | 161 | 164 | 167 | 57
Participants
  Asthenia: Any: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Asthenia: Any | 49 | 51 | 57 | 69 | 20
  Asthenia: Grade 3: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Asthenia: Grade 3 | 3 | 9 | 11 | 9 | 2
  Fever: Any: number analyzed (Participants) | 162 | 159 | 159 | 164 | 57
  Fever: Any | 5 | 8 | 8 | 5 | 1
  Fever: Grade 3: number analyzed (Participants) | 162 | 159 | 159 | 164 | 57
  Fever: Grade 3 | 0 | 0 | 1 | 0 | 0
  Headache: Any: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Headache: Any | 100 | 96 | 108 | 104 | 28
  Headache: Grade 3: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Headache: Grade 3 | 8 | 22 | 17 | 14 | 4
  Malaise: Any: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Malaise: Any | 72 | 75 | 97 | 90 | 26
  Malaise: Grade 3: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Malaise: Grade 3 | 10 | 17 | 19 | 13 | 3
  Myalgia: Any: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Myalgia: Any | 70 | 69 | 71 | 84 | 21
  Myalgia: Grade 3: number analyzed (Participants) | 162 | 160 | 159 | 164 | 57
  Myalgia: Grade 3 | 4 | 10 | 11 | 13 | 3

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to 28 days after each dose of CYD dengue vaccine or Placebo. Solicited Reaction (SR) data were collected within 7 and 14 days after each vaccination. Serious adverse event (SAE) data were collected throughout the study, up to 30 days post-vaccination 3 (up to Month 13).
Description: Analysis was performed on Safety Analysis Set.
Arm/Group | CYD Dengue Vaccine Phase III Lot 1 | CYD Dengue Vaccine Phase III Lot 2 | CYD Dengue Vaccine Phase III Lot 3 | CYD Dengue Vaccine Phase II Lot | Placebo
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/161 | 0/164 | 0/167 | 0/57
Serious Adverse Events (participants affected / at risk) | 10/163 | 9/161 | 5/164 | 9/167 | 1/57
Other Adverse Events (participants affected / at risk) | 136/163 | 131/161 | 135/164 | 140/167 | 41/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Phase III Lot 1 (N=163) | CYD Dengue Vaccine Phase III Lot 2 (N=161) | CYD Dengue Vaccine Phase III Lot 3 (N=164) | CYD Dengue Vaccine Phase II Lot (N=167) | Placebo (N=57)
Stress Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bartholin's Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign Body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypergammaglobulinaemia Benign Monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Calculus Ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Phase III Lot 1 (N=163) | CYD Dengue Vaccine Phase III Lot 2 (N=161) | CYD Dengue Vaccine Phase III Lot 3 (N=164) | CYD Dengue Vaccine Phase II Lot (N=167) | Placebo (N=57)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (3) | 4 (4) | 1 (4) | 3 (3)
Asthenia (General disorders) | 49 (66) | 51 (72) | 58 (74) | 69 (90) | 20 (26)
Injection Site Erythema (General disorders) | 22 (26) | 15 (20) | 25 (31) | 24 (32) | 0 (0)
Injection Site Haematoma (General disorders) | 12 (12) | 9 (11) | 12 (13) | 10 (10) | 6 (6)
Injection Site Pain (General disorders) | 73 (122) | 74 (114) | 73 (122) | 78 (122) | 11 (15)
Malaise (General disorders) | 72 (110) | 75 (116) | 97 (146) | 90 (126) | 26 (43)
Pyrexia (General disorders) | 6 (7) | 9 (11) | 9 (10) | 5 (6) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (13) | 6 (6) | 9 (11) | 8 (8) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 13 (13) | 14 (15) | 16 (18) | 14 (15) | 6 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 70 (100) | 69 (105) | 72 (111) | 84 (124) | 21 (30)
Headache (Nervous system disorders) | 103 (188) | 97 (186) | 108 (208) | 104 (201) | 28 (61)
Dysmenorrhoea (Reproductive system and breast disorders) | 7 (9) | 5 (9) | 2 (2) | 4 (5) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 3 (3) | 3 (3) | 6 (6) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 5 (5) | 7 (7) | 12 (13) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.